CLINICAL TRIAL: NCT05547087
Title: A Phase 2, Randomized, Double-Blind, Dose Finding Study to Describe the Immunogenicity, Safety and Tolerability of VN-0200 in Japanese Adults Aged 60-80 Years
Brief Title: A Dose Finding Study of VN-0200
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VN0200-091
Record Dates: First submitted 2022-09-15; First posted 2022-09-21 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Group 1: VN-0200 low dose (Experimental): Healthy elderly subjects will be randomized to receive intramuscular injection of low dose of VAGA-9001a.
  Interventions: Biological: VN-0200
- Group 2: VN-0200 low dose (Experimental): Healthy elderly subjects will be randomized to receive intramuscular injection of low dose of VAGA-9001a adjuvanted with low dose of MABH-9002b.
  Interventions: Biological: VN-0200
- Group 3: VN-0200 low dose (Experimental): Healthy elderly subjects will be randomized to receive intramuscular injection of low dose of VAGA-9001a adjuvanted with medium dose of MABH-9002b.
  Interventions: Biological: VN-0200
- Group 4: VN-0200 low dose (Experimental): Healthy elderly subjects will be randomized to receive intramuscular injection of low dose of VAGA-9001a adjuvanted with high dose of MABH-9002b.
  Interventions: Biological: VN-0200
- Group 5: VN-0200 medium dose (Experimental): Healthy elderly subjects will be randomized to receive intramuscular injection of medium dose of VAGA-9001a.
  Interventions: Biological: VN-0200
- Group 6: VN-0200 medium dose (Experimental): Healthy elderly subjects will be randomized to receive intramuscular injection of medium dose of VAGA-9001a adjuvanted with high dose of MABH-9002b.
  Interventions: Biological: VN-0200
- Group 7: VN-0200 high dose (Active Comparator): Healthy elderly subjects will be randomized to receive intramuscular injection of high dose of VAGA-9001a.
  Interventions: Biological: VN-0200
- Group 8: VN-0200 high dose (Experimental): Healthy elderly subjects will be randomized to receive intramuscular injection of high dose of VAGA-9001a adjuvanted with low dose of MABH-9002b.
  Interventions: Biological: VN-0200
- Group 9: VN-0200 high dose (Experimental): Healthy elderly subjects will be randomized to receive intramuscular injection of high dose of VAGA-9001a adjuvanted with medium dose of MABH-9002b.
  Interventions: Biological: VN-0200
- Group 10: VN-0200 high dose (Experimental): Healthy elderly subjects will be randomized to receive intramuscular injection of high dose of VAGA-9001a adjuvanted with high dose of MABH-9002b.
  Interventions: Biological: VN-0200

INTERVENTIONS:
Biological: VN-0200 — VN-0200 (antigen: VAGA-9001a, adjuvant: MABH-9002b) administered as an intramuscular injection; 2 shots in 4 weeks.

SUMMARY:
This study will assess the immunogenicity, safety and tolerability of VN-0200 after intramuscular injections in Japanese healthy elderly subjects.

ELIGIBILITY:
Inclusion Criteria:

* Japanese healthy elderly aged >=60 and =<80 years (at the time of informed consent).
* Subjects who can follow the compliance requirements during clinical trials, undergo medical examinations and tests specified by the protocol, and report symptoms, etc.

Exclusion Criteria:

* Serious cardiovascular, respiratory, hepatic, renal, gastrointestinal, or neuropsychiatric disorders.
* Serious acute illness.
* Has been diagnosed with congenital or acquired immunodeficiency.
* Previous vaccination with an RSV vaccine (including the investigational drugs).
* Having a history of anaphylaxis or severe allergies due to medicines, or vaccination.
* Administration of gamma globulins, systemic immunosuppressants (including drugs for the treatment of autoimmune diseases), hematopoietics (excluding iron and vitamins), and corticosteroids (excluding topical preparations, inhalants, and small-dose short-term oral administration*) or planned administration of them in the period starting 28 days prior to informed consent and ending 28 days after the second vaccination. * <14 days, 20 mg/day on a prednisolone basis.
* Planned or actual administration of other vaccine in the period starting 14 days prior to informed consent and ending 14 days after the second vaccination.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2022-10-13 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Geometric Mean Titer (GMT) of anti-RSV Subgroup A (RSV/A) Neutralizing Activity | Day 57 (28 days after the second dosing of the investigational product)
Geometric Mean Fold Rise (GMFR) of Anti-RSV/A Neutralizing Activity | Day 57 (28 days after the second dosing of the investigational product)

SECONDARY OUTCOMES:
Geometric Mean Titer (GMT) of Anti-RSV/A Neutralizing Activity | Day 29 (the second dosing of the investigational product)
Geometric Mean Fold Rise (GMFR) of Anti-RSV/A Neutralizing Activity | Day 29 (the second dosing of the investigational product)
Geometric Mean Titer (GMT) of Anti-RSV/B Neutralizing Activity | Day 29 (the second dosing of the investigational product) and Day 57 (28 days after the second dosing of the investigational product)
Geometric Mean Fold Rise (GMFR) of Anti-RSV/B Neutralizing Activity | Day 29 (the second dosing of the investigational product) and Day 57 (28 days after the second dosing of the investigational product)
Geometric Mean Titer (GMT) of Anti-VAGA-9001a Immunoglobulin G (IgG) | Day 29 (the second dosing of the investigational product) and Day 57 (28 days after the second dosing of the investigational product)
Geometric Mean Fold Rise (GMFR) of Anti-VAGA-9001a Immunoglobulin G (IgG) | Day 29 (the second dosing of the investigational product) and Day 57 (28 days after the second dosing of the investigational product)
VAGA-9001a Specific IFN-Gamma Production Responses | Day 29 (the second dosing of the investigational product) and Day 57 (28 days after the second dosing of the investigational product)
Number of Participants Reporting Solicited Adverse Events (Local and Systemic Adverse Reactions) and Side Reactions | Day 1 (the first dosing of the investigational product) up to Day 8, Day 29 (the second dosing of the investigational product) up to Day 36 and at time of discontinuation (whichever comes first), up to approximately 1 month
Number of Participants Reporting Non-Solicited Adverse Events and Side Reactions | Day 1 (the first dosing of the investigational product) up to Day 57 (28 days after second dosing of the investigational product) and at time of discontinuation (whichever comes first), up to approximately 2 months
Number of Participants Reporting Serious Adverse Events and Side Reactions | From date of informed consent up to approximately 12 months
Number of Participants Reporting Potential Immune-Mediated Disease | Day 1 (the first dosing of the investigational product) up to the time of follow-up and discontinuation (up to approximately 12 months)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Leader, Study Director — Daiichi Sankyo
Locations (3):
- Japan (3):
  - SOUSEIKAI PS Clinic, Hakata, Fukuoka
  - SOUSEIKAI Sumida Hopital, Sumida City, Tokyo
  - SOUSEIKAI Nishi-Kumamoto Hospital, Kumamoto

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/